CLINICAL TRIAL: NCT04592653
Title: Clinical and Immunologic Activity of Nemvaleukin Alfa With Less Frequent IV Dosing Schedule as Monotherapy and in Combination With Pembrolizumab and Impact on Tumor Microenvironment in Solid Tumor Patients - ARTISTRY-3
Brief Title: Less Frequent IV Dosing & Tumor Microenvironment (TME) Study of Nemvaleukin Alfa (ALKS 4230) Monotherapy and in Combination With Pembrolizumab (ARTISTRY-3)
Acronym: ARTISTRY-3
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mural Oncology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALKS 4230-003
Record Dates: First submitted 2020-08-24; First posted 2020-10-19 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumor
Keywords: Alkermes; IL-2; Interleukin-2; Oncology; Immuno-oncology; Cytokine; Pembrolizumab; Keytruda; PD-L1; Solid tumors; Immunotherapy; Nemvaleukin
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Tumor Microenvironment (TME) Nemvaleukin and Pembrolizumab (Experimental): Nemvaleukin will be administered via Intravenous (IV) infusion given daily for 5 consecutive days followed by an off-treatment period. Starting on Cycle 3, Day 1 of each cycle, Pembrolizumab will be administered via IV infusion followed by IV infusion of nemvaleukin
  Interventions: Biological: Nemvaleukin alfa; Biological: Pembrolizumab
- Cohort 2 Part A: Less Frequent IV Dosing Nemvaleukin (Experimental)
  Interventions: Biological: Nemvaleukin alfa
- Cohort 2 Part B: Less Frequent IV Dosing Nemvaleukin and Pembrolizumab (Experimental): This arm will not open for enrollment.
  Interventions: Biological: Nemvaleukin alfa; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Nemvaleukin alfa — IV infusion over 30 minutes
  Other Names: ALKS 4230
Biological: Pembrolizumab — IV infusion over 30 minutes
  Other Names: Keytruda
  Arms: Cohort 1: Tumor Microenvironment (TME) Nemvaleukin and Pembrolizumab; Cohort 2 Part B: Less Frequent IV Dosing Nemvaleukin and Pembrolizumab

SUMMARY:
The study will be conducted in 2 cohorts. A single-center design for the tumor microenvironment (TME) cohort (Cohort 1), and a multicenter design for the less frequent intravenous (IV) dosing cohort (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of an advanced solid tumor type of cutaneous melanoma, RCC, TNBC, MSS colorectal cancer, MSI-H solid tumors (NOS), or ovarian cancer with at least 1 accessible lesion for biopsy (Cohort 1 TME)
* Patients must have histologically or cytologically confirmed epithelial tumor of the fallopian tube, peritoneum, or ovaries, cervical cancer, endometrial cancer, non-small cell lung adenocarcinoma, small cell lung cancer, gastric and gastroesophageal junction adenocarcinoma, esophageal cancer (squamous and adeno cell type), pancreatic cancer, biliary tract tumor (including intra- and extrahepatic cholangiocarcinoma, gall bladder, ampullary type), cutaneous melanoma, mucosal melanoma, head and neck squamous cell carcinoma, or metastatic or advanced breast cancer after treatment failure or intolerance of 1 to 3 established indication specific therapies (Cohort 2)
* Patient must have received 1 to 3 prior FDA-approved targeted therapies, failure of adjuvant and neoadjuvant therapy is considered 1 line of treatment
* All patients' baseline biopsies must be taken no more than 3 months before Screening and at least 4 weeks after completion of last antineoplastic therapy
* Patients must have at least 1 lesion that qualifies as a target lesion
* Patients must have adequate hematologic reserve
* Patients must have adequate hepatic and renal function
* For Cohort 1 (TME) and Part A of Cohort 2 (less frequent IV dosing), treatment with prior immunotherapy is permitted unless the patient has previously experienced grade ≥3 autoimmune toxicity or drug-related toxicity requiring discontinuation. Patients in Part B of Cohort 2 (less frequent IV dosing) who received prior anti-PD-(L)1 for at least 3 months may enroll if they had a response of stable disease or better
* For Cohort 1 (TME), patients who have received prior anti-PD-1 directed therapy must wait at least 4 weeks from last dose of such therapy before the Screening biopsy is collected
* Women of childbearing potential (WOCBP) must have a negative pregnancy test
* Additional criteria may apply

Exclusion Criteria:

* Patients with active or symptomatic central nervous system metastases
* Patients who require pharmacologic doses of systemic corticosteroids (greater than 10 mg of prednisone daily or equivalent)
* Patients known to be positive for HIV and/or history of hepatitis B, or C infections or is known to be positive for hepatitis B antigen (HBsAg)/hepatitis B virus (HBV) DNA or hepatitis C antibody (Hep C Ab) or RNA.
* Patients with a known additional malignancy within 2 years of the start of Screening
* Patients who have received radiotherapy within the last 4 weeks before start of study treatment
* Patients who have received systemic immunomodulatory agents within 4 weeks or 5 half lives, whichever is shorter, before Cycle 1 Day 1,
* Patients who have received prior IL-2-based or IL-15-based soluble protein therapy at any time in the past are excluded
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in density (cell counts per mm2) of immune cell (including total T cells, CD8+ T cells, CD56+ cells and Treg cells) | From the time of the Patient's pre-treatment biopsy to the time of the Patient's on-treatment biopsy
  Changes in density (cell counts per mm2) of immune cell (including total T cells, CD8+ T cells, CD56+ cells and Treg cells) based on immunohistochemistry (IHC) and/or immunofluorescence (IF) in the TME between pretreatment and on-treatment (Cycle 2 Day 8) paired tumor biopsies
Changes in ratios (including T/Treg, CD8+/Treg, CD56+/Treg) based on immunohistochemistry (IHC) and/or immunofluorescence (IF) in the TME between pretreatment and on-treatment (Cycle 2 Day 8) paired tumor biopsies | From the time of the Patient's pre-treatment biopsy to the time of the Patient's on-treatment biopsy
Incidence of dose-limiting toxicity (DLT) | From the first dose through end of dose-limiting toxicity observation period (up to 24 months)

SECONDARY OUTCOMES:
Proportion of subjects with objective evidence of Complete or Partial Response [(CR)/immune CR (iCR) or (PR) immune PR (iPR)](CR)/immune CR (iCR) | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months
Duration of response in subjects with Complete or Partial Response [(CR)/immune CR (iCR) or (PR) immune PR (iPR)] | Time from the first documentation of complete response or partial response to the first documentation of objective tumor progression or death due to any cause (estimated up to 24 months)
Incidence of Adverse Events | Time from first dose of study drug to the end of study (estimated up to 24 months)
Incidence of drug-related Serious Adverse Events | Time from first dose of study drug to the end of study (estimated up to 24 months)
Incidence of drug-related Adverse Events leading to discontinuation | Time from first dose of study drug to the end of study (estimated up to 24 months)
Serum concentrations of ALKS 4230 | From time of initiation of therapy until the last treatment cycle (each cycle is 14 or 21 days), assessed up to 24 months
  Concentration data will be summarized by dose level
Serum will be assayed for the presence of anti-ALKS 4230 antibodies | From time of initiation of therapy until the last treatment cycle (each cycle is 14 or 21 days), assessed up to 24 months
  Results will be summarized by dose level
Changes in absolute cell numbers (including total T cells, CD8+ T cells, NK cells and Treg cells) | From time of initiation of therapy until the last treatment cycle (each cycle is 14 or 21 days), assessed up to 24 months
  Changes in absolute cell numbers (including total T cells, CD8+ T cells, NK cells and Treg cells) between pretreatment and on-treatment serial peripheral blood samples obtained from patients being treated with ALKS 4230 monotherapy and with the combination of ALKS 4230 plus pembrolizumab
Changes in ratios (including T/Treg, CD8+/Treg, NK/Treg) between pretreatment and on treatment | From time of initiation of therapy until the last treatment cycle (each cycle is 14 or 21 days), assessed up to 24 months
  Changes in ratios (including T/Treg, CD8+/Treg, NK/Treg) between pretreatment and on-treatment serial peripheral blood samples obtained from patients being treated with ALKS 4230 monotherapy and with the combination of ALKS 4230 plus pembrolizumab
Serum concentrations of proinflammatory cytokines, including IFNγ, TNF-α, IL-1B, IL-6, IL-10, will be assessed using a multiplex method from initiation of therapy | From time of initiation of therapy until the last treatment cycle (each cycle is 14 or 21 days), assessed up to 24 months
Changes in absolute numbers of circulating leukocytes | From time of initiation of therapy until the last treatment cycle (each cycle is 14 or 21 days), assessed up to 24 months
  Changes in absolute numbers of circulating leukocytes between pretreatment and on-treatment serial peripheral blood samples obtained from patients being treated with ALKS 4230 monotherapy and with the combination of ALKS 4230 plus pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Mural Oncology
Locations (6):
- United States (4):
  - START Midwest, Grand Rapids, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - START Mountain, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia
- Spain (2):
  - Hospital Clinico San Carlos, Madrid
  - CIOCC HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Undecided